CLINICAL TRIAL: NCT01784094
Title: Connective Tissue Motion Measure 2
Status: Completed | Type: Observational
Sponsor: Stromatec, Inc. (Industry)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Robert Davis, Principal Investigator, Stromatec, Inc.
Other Study IDs: 2R44AT006085 (NIH)
Record Dates: First submitted 2013-01-30; First posted 2013-02-05 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Low Back Pain; Musculoskeletal Pain
MeSH Terms: conditions — Low Back Pain; Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Low back pain subjects: Subjects with chronic or recurrent low back pain
  Interventions: Device: StromaGlide
- No low back pain subjects: Subjects who are generally healthy with no low back pain
  Interventions: Device: StromaGlide

INTERVENTIONS:
Device: StromaGlide

SUMMARY:
This study aims to compare the Connective Tissue Motion Measure (CTMM) in low back pain and no-low back pain subjects, evaluate the reliability of the CTMM, and examine the correlation of CTMM with low back pain symptoms, disability, and functional measures. The investigators hypothesize that CTMM will be reduced, on average, in low back pain subjects, that CTMM will be reliable with an intra-class correlation greater than 0.8, and CTMM will negatively correlate with low back pain symptoms, disability and functional measures.

ELIGIBILITY:
Inclusion Criteria for all subjects:

* able to stand and walk without assistance
* able to read and understand English
* able to understand and sign a consent form

Inclusion Criteria for low back pain subjects:

* history of recurrent or chronic low back pain

Inclusion criteria for no-low back pain subjects:

* no history of low back pain or other chronic pain that has limited activities of daily living or work
* numerical chronic pain index of less than 0.5

Exclusion Criteria for all subjects:

* previous severe back or lower extremity injury or surgery
* major structural spinal deformity (scoliosis, kyphosis, stenosis)
* ankylosing spondylitis or rheumatoid arthritis
* neurological deficit (weakness or sensory loss, decreased deep tendon reflexes suggesting nerve root compression, but not subjective symptoms of nerve root irritation (sciatica))
* radicular pain
* neurological or major psychiatric disorder
* bleeding disorders
* corticosteroid or anticoagulant medication
* substance abuse
* pregnancy
* active worker's compensation or disability case
* in litigation for a low back pain problem
* acute systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Connective Tissue Shear Strain Motion | Baseline
Change in Connective Tissue Shear Strain Motion | Baseline to 1 hour
Change in Connective Tissue Shear Strain Motion | Baseline to one day
Change in Connective Tissue Shear Strain Motion | Baseline to one week

CONTACTS AND LOCATIONS:
Locations (1):
- Stromatec, Inc, Burlington, Vermont, United States